CLINICAL TRIAL: NCT06146114
Title: Single Center Registration Study on HER2 Expression and Clinical Pathological Characteristics in Prostate Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: bks03
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: HER2 Expression and Clinical Pathological Characteristics in Prostate Cancer
Keywords: HER2; prostate cancer; clinical pathological characteristics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: 1. Prostate cancer patients confirmed by histopathology in our hospital from January 2018 to July 2023;
  2. Men aged ≥ 18 years old;
  3. The expected survival time is greater than 12 weeks;
  4. The KPS functional status score is greater than 60, and the ECOG status score is 0-2 points;
  5. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.
  Interventions: Diagnostic Test: Collect HER2 expression in prostate cancer patients

INTERVENTIONS:
Diagnostic Test: Collect HER2 expression in prostate cancer patients — HER2 testing and disease information collection for patients diagnosed with prostate cancer and able to obtain tumor tissue in our hospital from January 2018 to July 2023

SUMMARY:
This study is a single center, non-interference, retrospective registration study: HER2 testing and disease information collection were conducted on patients diagnosed with prostate cancer and able to obtain tumor tissue in our hospital from January 2018 to July 2023. Statistical analysis was conducted on the collected information to analyze the expression of HER2 in Chinese prostate patients and the correlation between HER2 and disease type.

DETAILED DESCRIPTION:
1. To explore the expression of HER2 protein in prostate cancer patients admitted to Qilu Hospital of Shandong University, especially the expression rate of HER2 protein under different pathological characteristics (age, TNM grade, primary and metastasis), and to explore the correlation between HER2 protein expression level, efficacy, and prognosis based on patient clinical information.
2. (1) Main Purpose

Analyze the expression of HER2 in prostate cancer patients admitted to Qilu Hospital of Shandong University.

(2) Secondary purpose

The expression of HER2 protein under different clinical and pathological characteristics (age, TNM grade, primary, and metastasis).

3.Main indicators:

The expression of HER2 in prostate cancer patients.

Secondary indicators:

1. The correlation between HER2 expression (IHC0/1+/2+/3+) and disease characteristics in locally advanced or metastatic prostate cancer patients;
2. The distribution of HER2 expression in different ages, different parts, different degrees of differentiation, and different TNM stages; Evaluate the expression of primary and metastatic lesions in patients with metastasis

ELIGIBILITY:
Inclusion Criteria:

* 1. Prostate cancer patients confirmed by histopathology in our hospital from January 2018 to July 2023;

  2. Men aged ≥ 18 years old;

  3. The expected survival time is greater than 12 weeks;

  4. The KPS functional status score is greater than 60, and the ECOG status score is 0-2 points;

  5. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

- 1. Those who have been diagnosed with tumors in other parts, such as lung cancer, liver cancer, stomach cancer, colorectal cancer, breast cancer, etc. (except for cancer in situ or non melanoma skin cancer, or combined tumors with low recurrence probability within a few years);

2. According to the researcher's judgment, there are other patients who are not suitable for inclusion.

Ages: 50 Years to 90 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: HER2 testing and disease information collection for patients diagnosed with prostate cancer and able to obtain tumor tissue in our hospital from January 2018 to July 2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
HER2 expression in prostate cancer patients | 18 months
  HER2 test results

SECONDARY OUTCOMES:
Correlation between HER2 expression (IHC0/1+/2+/3+) and disease characteristics in locally advanced or metastatic prostate cancer patients | 18 months
The distribution of HER2 expression in different ages, different parts, different degrees of differentiation, and different TNM stages; | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No